CLINICAL TRIAL: NCT03351634
Title: EVALUATION OF THE SAFETY AND EFFICACY OF ADJUSTABLE CONTINENT THERAPY FOR THE MANAGEMENT OF NEUROGENIC INCONTINENCE IN CHILDREN WITH SPINAL DYSRAPHISM.
Brief Title: EVALUATION OF THE SAFETY AND EFFICACY OF ADJUSTABLE CONTINENT THERAPY IN CHILDREN WITH SPINAL DYSRAPHISM.
Acronym: BPUA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-49; 2016-A01974-47 (Registry Identifier: ANSM)
Record Dates: First submitted 2017-08-25; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Neurogenic Bladder Due to Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with neurogenic incontinence with spinal dysraphism (Experimental)
  Interventions: Device: Implantation of ACT balloon, Uromedica (Irvine, CA, USA) periurethrally at the bladder neck

INTERVENTIONS:
Device: Implantation of ACT balloon, Uromedica (Irvine, CA, USA) periurethrally at the bladder neck — The ACT system is a permanent implant designed for the correction of incontinence in patients.

SUMMARY:
Urinary continence is still a difficult goal to achieve in neurogenic bladder patients. Conservative treatment of neurogenic urinary incontinence using clean intermittent catheterization in conjunction with pharmacological therapy, notably anticholinergic medication +/- adrenergic agents, may produce continence in a variable number of patients. In other patients, reconstructive surgery of the bladder and/or bladder neck is necessary to achieve urinary continence. Surgical treatment options to increase bladder outlet resistance in patients with neurogenic bladder include injection of bulking agents around the bladder neck, bladder neck reconstruction, fascial sling procedures and Artificial Urinary Sphincter.

The Adjustable Continence Therapy system (ACT) or periurethral adjustable balloons are a minimally invasive device consisting of two volume-adjustable balloons implanted periurethrally at the bladder neck as a method of augmenting titration for urethral coaptation. Adjustable means that such system would be adaptable to the individual clinical condition.

Originally conceived and developed as a treatment for female stress urinary incontinence, the technique has been then adapted and balloons were globally developed for the use in postprostatectomy incontinence. The published success rate in male after prostatectomy and in women was respectively 56 to 92% and 60 to 83%.

The investigators hypothesize that the use of ACT for treating incontinence in children secondary to neurogenic sphincter incontinence could compress the urethra or the bladder neck, acting as an extrinsic occlusive system increasing passive and dynamic urethral and bladder resistance.

Goal of the study:

To prospectively assess the efficacy and safety of periurethral adjustable balloons in the treatment of neurogenic incontinence in children with spinal dysraphism.

Material and methods :

A prospective study will be performed at La Timone Enfants hospital and La Nord hospital in Marseille, France. Boys and girls at least at school age (5 or 6 years) with neurogenic incontinence due to outlet issues (low detrusor leak point pressure and low stress leak point pressure) with spinal dysraphism will be recruited.

The ACT balloon is an implantable medical device developed and furnished for free by Uromedica (Irvine, CA, USA). The procedure is performed under general anaesthesia using the same implantation technique as published in adult population.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls > 5 years with spinal dysraphism (occult or open)
* Neurogenic sphincteric incontinence (leak point pressure < 45 cm d'H20, open bladder neck during filling, urinary incontinence)
* Normal renal function (eGFR > 90ml/min)
* No (or stable) upper urinary tract dilatation in ultrasound
* In case no compliante bladder ( bladder capacity < 50% for the age) a concomitant injection of botox endoscopically will be performed

Exclusion Criteria:

* under 5 years with an acquired neurogenic bladder
* renal insufficiency (acute or chronic)
* evolutive deterioration of the upper urinary tract (hydronephrosis)
* active systemic or urinary tract infections
* unmanageable detrusor instability
* reduced bladder compliance
* residual volume greater than 100 ml after voiding
* bleeding disorders
* urethral stenosis
* who refused CIC
* patent sacral bedsore

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of urinary continence with the Schulte-Baukloh score and 24hours pad-test | 5 YEARS
  Evaluation of urinary continence with mictional schedule and 24hours pad-test (Patients will be classified as "dry" if they will be using no pads or a single ''security pad'' per day; "significantly improved" if a reduction >50% in pad usage (usually representing 2- 5 pads/day, depending on preoperative pad use); and little/no improvement (>5 pads/day and <50% improvement against baseline) and the Schulte-Baukloh score

SECONDARY OUTCOMES:
Evaluation of the quality of life with the PIN-Q score | 5 YEARS
  The child will be asked to answer some items

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — ASSISTANTE PUBLIQUE HOPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France